CLINICAL TRIAL: NCT06059638
Title: BradycArdia paCemaKer With AV Interval Modulation for Blood prEssure treAtmenT
Acronym: BACKBEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orchestra BioMed, Inc (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS-08
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; Hypertension, Systolic; Hypertension, Essential
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): AVIM therapy activated with continued stable antihypertensive drug therapy
  Interventions: Device: Medtronic Astra/Azure DR MRI IPG with AVIM therapy Activated
- Control Group (Sham Comparator): AVIM therapy deactivated with continued stable antihypertensive drug therapy
  Interventions: Device: Medtronic Astra/Azure DR MRI IPG with AVIM therapy Deactivated

INTERVENTIONS:
Device: Medtronic Astra/Azure DR MRI IPG with AVIM therapy Activated — Antihypertensive therapy utilizing atrioventricular interval modulation.
  Other Names: BackBeat CNT
  Arms: Treatment Group
Device: Medtronic Astra/Azure DR MRI IPG with AVIM therapy Deactivated — AVIM therapy is deactivated
  Arms: Control Group

SUMMARY:
A prospective, multinational, randomized, double-blind, clinical trial evaluating the safety and effectiveness of a novel atrioventricular interval modulation (AVIM) algorithm downloaded into a dual-chamber Medtronic Astra/Azure pacemaker.

DETAILED DESCRIPTION:
The study will be conducted in three phases: 1) Screening Phase, 2) Double-blind Randomized Phase (1 year), and 3) Unblinded Phase (2 years). Patients scheduled for implantation of an Astra/Azure pacemaker, or those who already have one implanted, who also have hypertension, may be screened for inclusion into this study. Subjects meeting randomization eligibility criteria will have the investigational AVIM Therapy RAMware downloaded into the Astra/Azure pacemaker and be randomized 1:1 to either have AVIM therapy turned ON or turned OFF. All subjects will continue to receive antihypertensive drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has or is indicated for a dual-chamber pacemaker. Visit 1 can be performed within 30 days prior to a planned implant of a Medtronic Astra/Azure dual-chamber pacemaker system or at any time thereafter
2. On a stable antihypertension treatment regimen with at least 1 class of antihypertensive drug
3. Office SBP ≥135 mmHg and <180 mmHg
4. Average 24-Hour aSBP ≥130 mmHg and <170 mmHg

Exclusion Criteria:

1. LVEF <50%
2. NYHA Class III-IV
3. History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months
4. Myocardial infarction (MI) within 3 months
5. Prior percutaneous or surgical coronary, carotid, or endovascular intervention within 3 months
6. Permanent atrial fibrillation
7. Mitral valve regurgitation greater than or equal to grade 3
8. Aortic stenosis with a valve area less than 1.5 cm2
9. Has an active or prior device-based anti-hypertensive treatment (e.g., renal denervation procedure, baroreflex activation therapy)
10. Has an existing active cardiac device or neurostimulator other than the recent Astra/Azure pacemaker implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean 24-hour ambulatory systolic blood pressure (aSBP) at 3 Months | Baseline and 3 months post randomization
  Between group difference in the change of mean 24-hour ambulatory systolic blood pressure (aSBP) from baseline to 3 months post randomization
Freedom from Unanticipated Serious Adverse Device Effects (USADE) | 3 months post randomization
  Freedom from Unanticipated Serious Adverse Device Effects (USADE) in the treatment group at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute; Andrea Russo, MD, Principal Investigator — Cooper University
Locations (94):
- United States (66):
  - HonorHealth, Scottsdale, Arizona
  - Adventist Health Glendale, Glendale, California
  - Stanford, Redwood City, California
  - Scripps Clinic, San Diego, California
  - Sutter Valley Hospitals, San Francisco, California
  - South Denver Cardiology, Denver, Colorado
  - Intermountain Health Lutheran Hospital, Golden, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - HCA Florida JFK Hospital, Atlantis, Florida
  - Cardiovascular Research Solutions (MyCardiologist), Celebration, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Citrus Cardiology Consultants, Crystal River, Florida
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Baptist Health Jacksonville, Jacksonville, Florida
  - Baptist Health South Florida, Miami, Florida
  - Mount Sinai Medical Center of Florida, Miami Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - Wellstar Research Institute, Marietta, Georgia
  - St. Luke's Idaho Cardiology, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - West Houston Area Clinical Trial Consultants (Wichita, KS), Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - UMH-Sparrow Clinical Research, Lansing, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Health Partners Institute (Methodist Heart and Vascular Center), Bloomington, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St. Louis, St Louis, Missouri
  - The Cooper Health System, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virtua Medical Group, P.A., Marlton, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Lovelace Medical Center (New Mexico Heart Institute), Albuquerque, New Mexico
  - Northwell Health, Inc., New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - HCA Asheville Cardiology Associates, Asheville, North Carolina
  - Atrium Health - Sanger Heart, Charlotte, North Carolina
  - WakeMed, Raleigh, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - OhioHealth Corporation, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Hightower Clinical Trials, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Penn Medicine Lancaster General Health, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Ascension St. Thomas Hospital, Nashville, Tennessee
  - Ascension Seton, Austin, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Centra Health dba Stroobants Cardiovascular Center, Lynchburg, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Advocate Aurora Research Institute, LLC, Milwaukee, Wisconsin
- Belgium (5):
  - OLV Ziekenhuis, Aalst
  - Middelheim Ziekenhuis, Antwerp
  - Universite Libre de Bruxelles-Erasme Hospital, Brussels
  - UZ Brussel, Brussels
  - UZ Leuven, Leuven
- Czechia (2):
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
  - Na Homolce Hospital, Prague
- Germany (4):
  - Cardioangiologisches Centrum Bethanien (CCB) am AGAPLESION Markus Krankenhaus, Frankfurt
  - University Medical Centre Mannheim, Mannheim
  - Saarland University Hospital, Saarbrücken
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- Hungary (2):
  - Semmelweis University, Budapest
  - University of Debrecen, Debrecen
- Netherlands (2):
  - Amsterdam University Medical Centre, Amsterdam
  - Maastricht UMC+, Maastricht
- Poland (4):
  - Jagiellonian University Hospital, Krakow
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Silesian Center for Heart Diseases, Zabrze
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínico de Barcelona, Barcelona
  - La Paz University Hospital, Madrid
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
- United Kingdom (5):
  - Royal Brompton, London
  - St. Bartholomew's Hospital, London
  - St. Thomas Hospital, London
  - John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalarus Z, Merkely B, Neuzil P, Grabowski M, Mitkowski P, Marinskis G, Erglis A, Kazmierczak J, Sturmberger T, Sokal A, Pluta S, Geller L, Osztheimer I, Malek F, Kolodzinska A, Mika Y, Evans SJ, Hastings HM, Burkhoff D, Kuck KH. Pacemaker-Based Cardiac Neuromodulation Therapy in Patients With Hypertension: A Pilot Study. J Am Heart Assoc. 2021 Aug 17;10(16):e020492. doi: 10.1161/JAHA.120.020492. Epub 2021 Aug 13. PMID 34387126
- [Background] Neuzil P, Merkely B, Erglis A, Marinskis G, de Groot JR, Schmidinger H, Rodriguez Venegas M, Voskuil M, Sturmberger T, Petru J, Jongejan N, Aichinger J, Kamzola G, Aidietis A, Geller L, Mraz T, Osztheimer I, Mika Y, Evans S, Burkhoff D, Kuck KH; BackBeat Study Investigators. Pacemaker-Mediated Programmable Hypertension Control Therapy. J Am Heart Assoc. 2017 Dec 23;6(12):e006974. doi: 10.1161/JAHA.117.006974. PMID 29275370